CLINICAL TRIAL: NCT01587625
Title: High Dose Versus Low Dose Oxytocin for Augmentation of Delayed Labour
Acronym: OxyHighLow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Oxytocin high low dose
Record Dates: First submitted 2012-04-19; First posted 2012-04-30 (Estimated); Last update posted 2019-03-04 (Actual); Status verified 2019-03

CONDITIONS: Birth; Delayed
Keywords: Delayed labour; dystocia; oxytocin augmentation; primiparous women; childbirth; childbirth experience; progress
MeSH Terms: conditions — Dystocia | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High dose of oxytocin infusion (Experimental): Oxytocin: High dose infusion
  Interventions: Drug: Oxytocin
- Low dose of oxytocin infusion (Active Comparator): Oxytocin: Low dose infusion
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin

SUMMARY:
In a randomized control trial conducted in six study centers/labour wards in Sweden, consenting nulliparous women in active phase of labour and with a defined delayed labour progress will be randomized to receive a regimen of either high or low dose of oxytocin. Primary outcome is caesarean delivery rate. Secondary outcomes are: Apgar score, need of neonatal intensive care, hyper-stimulation of contractions, spontaneous vaginal birth rate, length of labour, postpartum haemorrhage, sphincter lacerations, experienced labour pain, epidural analgesia and the women´s childbirth experience one month postpartum (assessed with Childbirth Experience Questionnaire). Study results will contribute to establish good evidence-based routines regarding oxytocin treatment of delayed labour progress.

DETAILED DESCRIPTION:
The aim is to compare starting dose and increment of amount of oxytocin for augmentation of delayed labour to determine whether augmentation by high dose of oxytocin improves labour outcomes compared with a low dose of oxytocin, without effecting neonatal outcomes or birth experiences negatively.

Delay in labour, also described as poor progress, due to ineffective uterine contraction is a major problem in modern obstetric care and one of the main reasons for the increased rate of caesarean deliveries, in particular among nulliparous women. Infusion with synthetic oxytocin is a commonly used treatment of hypotonic uterine contractions. Despite the widespread use of oxytocin no consensus exists regarding the dosage of oxytocin, both starting dose and increment of amount of oxytocin.

In a randomized control trial conducted in six study centers/labour wards in Sweden, consenting nulliparous women in active phase of labour and with a defined delayed labour progress will be randomized to receive a regimen of either high or low dose of oxytocin. The expected outcome is a decreased caesarean section rate and increased rate of spontaneous vaginal delivery for women with high dose of oxytocin for augmentation, without affecting neonatal outcomes or childbirth experiences negatively.

Primary outcome is caesarean delivery rate. Secondary outcomes are Apgar score, need of neonatal intensive care, hyper-stimulation of contractions, spontaneous vaginal birth rate, length of labour, postpartum haemorrhage, sphincter lacerations, experienced labour pain, epidural analgesia and the women´s childbirth experience one month postpartum (assessed with Childbirth Experience Questionnaire). Based on a sample size calculation (α=0.05, β=0.80), 1045 women will be needed in each group. Analysis will be performed by the intention to treat.

Study results will contribute to establish good evidence-based routines regarding oxytocin treatment of delayed labour progress.

ELIGIBILITY:
Inclusion Criteria:

* Healthy nulliparous women
* singleton pregnancy
* normal pregnancy
* cephalic presentation
* spontaneous onset of active labour
* at term (37 - 42weeks gestation)
* delay or arrest of active labour

Exclusion Criteria:

* Non-Swedish speaking women
* previous uterine surgery
* intrauterine growth retardation > - 22%
* malpresentation at time of inclusion
* intrapartal hemorrhage at time of inclusion
* nonreassuring fetal-heart pattern at time of inclusion
* meconium at time of inclusion

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1376 (Actual)
Dates: Start 2013-08; Primary Completion 2016-06-09 (Actual); Study Completion 2016-10-08 (Actual)

PRIMARY OUTCOMES:
Caesarean delivery rate | At birth
  data from clinical records

SECONDARY OUTCOMES:
Spontaneous vaginal birth rate | At birth
  data from clinical records
Length of labour | At birth
  data from clinical records
Hyper-stimulation of contractions | At birth
  data from clinical records
Postpartum haemorrhage | Two hours postpartum
  data from clinical records
Sphincter lacerations | At birth
  data from clinical records
Epidural analgesia | At birth
  data from clinical records
Experienced labour pain | Two hours postpartum
  VAS 0-100 mm where 100 is highest pain level
Childbirth experience | 1 month postpartum
  Childbirth Experience Questionnaire (CEQ)
Apgar score | Five minutes postpartum
  data from clinical records
Neonatal intensive care | 1 month postpartum
  data from clinical records

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Sahlgrenska University Hospital, Gothenburg
  - NU Hospital Group, Trollhättan

IPD SHARING:
Plan to Share IPD: Yes
Data for primary and secondary outcome measures from the two groups will be submitted to the Swedish National Data Service (Svensk Nationell Datatjänst, SND), a national authority responsible for administrating sharing of research data.

REFERENCES:
- [Derived] Selin L, Berg M, Wennerholm UB, Dencker A. Dosage of oxytocin for augmentation of labor and women's childbirth experiences: A randomized controlled trial. Acta Obstet Gynecol Scand. 2021 May;100(5):971-978. doi: 10.1111/aogs.14042. Epub 2021 Jan 28. PMID 33176392
- [Derived] Selin L, Wennerholm UB, Jonsson M, Dencker A, Wallin G, Wiberg-Itzel E, Almstrom E, Petzold M, Berg M. High-dose versus low-dose of oxytocin for labour augmentation: a randomised controlled trial. Women Birth. 2019 Aug;32(4):356-363. doi: 10.1016/j.wombi.2018.09.002. Epub 2018 Oct 16. PMID 30341003